CLINICAL TRIAL: NCT07043673
Title: Plasma Concentrations of the Non-protein-bound Form of Vancomycin in Intensive Care
Brief Title: Plasma Concentrations of the Non-protein-bound Form of Vancomycin
Acronym: FREEVANCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/058/OB; N° IDRCB : 2022-A00706-37 (Other: ANSM)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Plasma Concentration
Keywords: vancomycine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — whole blood from samples taken as part of routine care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vancomycin plasma dosage group: Any intensive care patient at the Rouen University Hospital undergoing a plasma vancomycin dosage carried out as part of routine care for a suspected or proven Gram + Cocci infection

SUMMARY:
In routine practice, the use of vancomycin must be accompanied by plasma concentration monitoring to ensure that pharmacodynamic targets are met and that plasma concentrations are not in toxic ranges.

Because vancomycin has high plasma protein binding and a free fraction exhibits marked inter-individual variability, this variability is increased in intensive care, monitoring is all the more imperative.

The factors influencing the concentration and/or free fraction of vancomycin are numerous and vary from one study to another. The striking fact of this work is that the link between the concentration of the total form and the concentration of the free form has not been established.

However, only plasma measurements of the total form of vancomycin are currently available to clinicians in routine practice, while only the free fraction is biologically active, responsible for its efficacy, but also for its toxicity in the event of an overdose. This paradox is widely highlighted by authors who have studied the free fraction of vancomycin, emphasizing the importance of continuing scientific research on this subject. Moreover, these studies are few in number, particularly in intensive care units, and their sample size is small, and they present biases, particularly those related to their essentially retrospective nature.

The failure to consider the free concentration of vancomycin in the therapeutic monitoring strategy is primarily explained by the fact that clinicians do not have access to plasma concentrations of the free form of drugs in routine practice. Thus, the guidelines do not include pharmacodynamic targets for the free concentration, due to the lack of scientific data on the subject.

DETAILED DESCRIPTION:
Since 2019, the Rouen University Hospital Pharmacology Laboratory has been measuring the non-protein-bound plasma concentrations of certain beta-lactam antibiotics. The analyzed sample comes from ultrafiltration of the plasma sample, a pre-analytical technique used in several studies on the free form of vancomycin. Access to this new technique at Rouen University Hospital gives us the opportunity to study free vancomycin concentrations in ICU patients.

This study therefore aims to investigate free vancomycin plasma concentrations in patients admitted to the ICU treated for suspected or proven Gram-positive cocci infection, and for whom a dosage has been prescribed as part of routine practice.

This prospective study aims to specifically analyze the concentration of the free form of vancomycin, but also to determine whether certain clinical or biological factors could predict this concentration. The long-term objective would be to be able to better individualize dosage regimens for vancomycin, a molecule with high inter-individual variability in intensive care patients, with the aim of reducing both underdoses, which are responsible for therapeutic failures, and overdoses, which are responsible for toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized in intensive care,
* Treated with vancomycin for a proven or suspected Gram-positive cocci infection,
* For whom a plasma vancomycin dose has been prescribed
* Patient who has been informed and has expressed verbal non-opposition. If the patient is unable to express their non-opposition (emergency situations), non-opposition must be obtained from the patient's representative, their trusted person, or, failing that, a relative.

Exclusion Criteria:

* Objection from the patient or their relatives
* Discontinuous administration of vancomycin
* Total plasma vancomycin levels measured 5 days or more prior to inclusion, with the plasma sample being stored in the laboratory for only 5 days, as is standard practice.
* Individuals not covered by a social security scheme
* Failure to perform the prescribed vancomycin dosage: discontinuation of vancomycin, death, etc.
* Vancomycin serum sample taken before the 24th hour, including the loading dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns any intensive care patient at the Rouen University Hospital undergoing a plasma vancomycin dosage carried out as part of routine care for a suspected or proven Gram + cocci infection.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Measurement of plasma concentration of the free form of vancomycin | 24 hours after the start of continuous vancomycin infusion treatment
  The primary endpoint is determined by the measurement of the plasma concentration of the free form of vancomycin during the total plasma concentration measurement after at least 24 hours of continuous infusion treatment.

SECONDARY OUTCOMES:
Measurement of the fraction of the non-protein-bound form of vancomycin in plasma | 24 hours
  The fraction unbound to plasma proteins (free form) of vancomycin will be determined by the ratio of the concentration of the free form to that of the total form, and expressed as a %.
To determine the areas under the 24-hour curve (AUC24h) for total plasma protein-bound forms of vancomycin | 24 hours
  The area under the 24-hour plasma concentration curve (AUC24h) is calculated for vancomycin by the product of the plasma concentration times 24, due to continuous administration. It is expressed in mg.h/L.
To compare the areas under the 24-hour curve (AUC24h) for total and non-plasma protein-bound forms of vancomycin | 24 hours
  The area under the 24-hour plasma concentration curve (AUC24h) is calculated for vancomycin by the product of the plasma concentration times 24, due to continuous administration. It is expressed in mg.h/L.
To determine the areas under the 24-hour curve (AUC24h) for non-plasma protein-bound forms of vancomycin | 24 hours
  The area under the 24-hour plasma concentration curve (AUC24h) is calculated for vancomycin by the product of the plasma concentration times 24, due to continuous administration. It is expressed in mg.h/L.
To assess the frequency of achieving vancomycin pharmacodynamic targets for its total plasma concentration | 24 hours
  The pharmacodynamic objective of vancomycin will be considered to be achieved when the AUC24h/MIC of the total form is greater than or equal to 400, corresponding to a total vancomycinemia greater than 17 mg/L, for the treatment of a Staphylococcus sp with a MIC of 1 mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PG GOUIN, Professor, Study Director — University Hospital, Rouen
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.